CLINICAL TRIAL: NCT03164148
Title: A Study to Observe the Change of the Biological Signal (Heart Rate) During the Combined Pituitary Stimulation Test
Brief Title: Heart Rate Variability (HRV) in Pituitary Adenoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Dong Jun Lim, Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KC17OESI0205
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case Evaluation by T-REX TRI00A (Experimental): Case evaluation consists of confirmation of hospital visit dates, any side effects of device, T-REX TRI00A
  Interventions: Device: T-REX TRI00A

INTERVENTIONS:
Device: T-REX TRI00A — Case management consists of confirmation of hospital visit date, checking the adverse effect

SUMMARY:
Several studies have been reported that heart rate is known to be associated with prognosis in chronic diseases and acute diseases. For example, a decrease in heart rate following myocardial infarction may lead to a higher mortality rate. It is also known to predict heart failure, diabetic neuropathy, and even depression.

The combined pituitary function test artificially induces hypoglycemia to observe the secretion of pituitary hormone. The degree of change in heart rate during hypoglycemia can predict the adequacy of the test, and heart rate can be changed according to the characteristic of the tumor. Also, the prognosis can be predicted based on this.

In our study, we used a licensed device approved by KFDA (Korea Food and Drug Administration) to measure heart rate variability in patients with pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 year old
* Those with Normal blood pressure range:

  90mmHg <systolic <140mmHg, 60mmHg <diastolic <100mmHg
* Voluntary participants who visited Seoul St. Mary's Hospital

Exclusion Criteria:

* Those who have been diagnosed with sleep disorders, diabetes, arrhythmia, psychiatric disorder, physical or mental breakdown, drug addicts
* Diabetes, hypertension, cardiovascular disease diagnosed by taking a drug related to the disease
* Pregnant or lactating women
* Those who drank within 12 hours before participating in the trial
* Those who are deemed inappropriate by clinical trial researchers

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-10-16 (Estimated); Study Completion 2018-05-16 (Estimated)

PRIMARY OUTCOMES:
Changes in Heart rate variability according to the types of pituitary adenoma | 5 month of initial recruit

CONTACTS AND LOCATIONS:
Overall Officials: DongJun Lim, M.D, PhD., Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided